CLINICAL TRIAL: NCT00074893
Title: Shock Absorbing Brace for Study of Upper Extremity Musculoskeletal Disorders
Brief Title: Protective Brace to Prevent Hand and Arm Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: NIAMS-079; 1R43AR049167-01 (NIH)
Record Dates: First submitted 2003-12-23; First posted 2003-12-24 (Estimated); Last update posted 2006-03-08 (Estimated); Status verified 2006-03

CONDITIONS: Cumulative Trauma Disorders; Carpal Tunnel Syndrome
Keywords: Repetitive Strain Injuries; Vibration Damping; Protective Brace; Piezoelectric; SmartWear
MeSH Terms: conditions — Cumulative Trauma Disorders; Carpal Tunnel Syndrome

INTERVENTIONS:
Device: piezoelectric wrist brace

SUMMARY:
When people use hand-held power tools, their hands and arms vibrate along with the tool they are holding. People who frequently use hand-held power tools may develop injuries related to this vibration. This study will evaluate a protective brace designed to prevent vibration-related hand and arms injuries.

DETAILED DESCRIPTION:
Workers who use hand-held power tools absorb significant vibration energy in their arms and hands and may develop musculoskeletal disorders (MSDs) such as carpal tunnel syndrome and hand-arm vibration syndrome. Protective braces may be worn to decrease the incidence of occupational MSDs. The National Institute for Occupational Safety and Health has identified key attributes for protective braces; these attributes include vibration damping, comfort, non-interference with worker dexterity, and maintenance of safe hand temperature. Most currently available braces do not adequately address these NIOSH requirements. This study will evaluate the efficacy of a brace with piezoelectric damping material.

Participants in the study will be fitted with a brace on each hand. One brace will have piezoelectric damping material and the other will be a currently available, off-the-shelf commercial brace. Hand-held joysticks and handles mounted to a vibration shaker table will be used to simulate power tool use. Participants will undergo a series of tests designed to measure hand acceleration and vibration while grasping the study joysticks and handles. The tests will take approximately 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Normal hand anatomy and full range of motion

Exclusion Criteria:

* History of significant hand or wrist arthritis
* Open wounds
* Prior hand or wrist surgery
* Neuropathies
* Skin hypersensitivity
* Contact dermatitis
* Reflex sympathetic dystrophy

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15
Dates: Start 2003-11; Study Completion 2004-02

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Pottenger, PhD, Principal Investigator — SmartWear, LLC
Locations (1):
- UCLA Hand Center, Los Angeles, California, United States